CLINICAL TRIAL: NCT06828458
Title: Determining Elements of Anti-Fungal Immunity in BURN Patients
Acronym: DEFI-BURN
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241672
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Burn
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood Rectal swab skin swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with burn injury
  Interventions: Other: Biological sampling

INTERVENTIONS:
Other: Biological sampling — Whole blood on EDTA sample 2 tubes (5mL) PAXgene sample 1 tube (2.5 mL) Rectal swab Skin swab (1 swab for 5 anatomically burned sites)
  At day 0, day 3, day 7, day 14, day 21

SUMMARY:
Scientific justification Invasive fungal diseases (IFDs) pose a substantial threat, especially in immunocompromised patients, necessitating urgent research focus and therapeutic advancements. The IFI-BURN study, involving a cohort of patients with severe burn injury (n=276), revealed a significant IFD incidence of 31.6% and underscored their critical impact on morbidity and mortality. While fungi are present everywhere, for moulds within the environment and for yeasts within our microbiota, why certain patients develop IFDs and others do not, remains poorly understood. The answer most likely resides in the impact of the burn injury on the immune response, loss of skin barrier and particular predisposing immune phenotype of patients. The immune system is composed of both cellular and humoral components, but the latter is far less studied in antifungal immunity although they exert multiple antimicrobial mechanisms.

ELIGIBILITY:
Inclusion Criteria:

Burn patients

* Adult patients ≥ 18 years old
* Admission < 4 days following burn injury
* Total burn surface Area ≥ 15%
* Non opposition of the patient or his/her relatives to the research
* Affiliation to social security or any health insurance

Exclusion Criteria:

* Pregnancy
* Opposition of the patient or his/her relatives
* Decision not to resuscitate or to limit or stop active therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with burn injury
Sampling Method: Non-Probability Sample
Enrollment: 327 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Invasive fungal disease (IFD) onset during hospitalisation time | Up to 18 months
  Proven IFD according to EORTC/MSGERC criteria applicable for invasive candidiasis. Putative invasive mold infection is defined with ≥ 2 positive culture from skin biopsy/bronchoalveolar lavage or ≥ 2 positive blood specific qPCR (aspergilosis, mucorales, fusariosis) or a combination of both. Possible invasive mold infection is defined with only one positive mycological criterion.

SECONDARY OUTCOMES:
Overall survival | At day 30
Overall survival | At day 90
Hospital mortality | Up to 18 months
Incidence of organ failure during hospitalisation | Up to 18 months
  * Acute respiratory distress syndrome defined by the modified Berlin criteria, or
  * Acute kidney injury as defined by the KDIGO consensus, or
  * Septic shock and doses of catecholamines defined by SEPSIS-3
Severity score at admission | At inclusion
  SAPS 2 : Simplified Acute Physiology Score II The score can range from 0 to 163. Higher score indicates more severe illness and a higher risk of mortality. Lower score indicates less severe illness and a lower risk of mortality.
Severity score at admission | At inclusion
  ABSI Acute Bowel Ischemia Severity Index The score ranges from 0 to 10. A higher score indicates a more severe case and a higher risk of mortality.
Severity score at admission | At inclusion
  SOFA score : Sequential Organ Failure Assessment The score can range from 0 to 24, with higher scores indicating more severe organ failure and a worse prognosis.
Number of days without renal replacement therapy | At day 30
Number of days without mechanical ventilation | At day 30
Length of stay in Intensive Care Unit | Up to 18 months
Length of stay in hospital | Up to 18 months

IPD SHARING:
Plan to Share IPD: Undecided